CLINICAL TRIAL: NCT00315575
Title: BOLD and Perfusion fMRI of Alzheimer's Disease Risk
Brief Title: Memory Imaging of Normal Aging
Status: Completed | Type: Observational
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Adam Fleisher, MD, University of California, San Diego
Other Study IDs: IA0092; 5K23AG024062-02 (NIH)
Record Dates: First submitted 2006-04-14; First posted 2006-04-18 (Estimated); Last update posted 2009-01-26 (Estimated); Status verified 2009-01

CONDITIONS: Alzheimer's Disease
Keywords: Dementia; brain circulation; disease /disorder proneness /risk; neuropathology; neurophysiology; aging; apolipoprotein E; genotype; hemodynamics; memory; temporal lobe /cortex
MeSH Terms: conditions — Alzheimer Disease; Dementia; Disease Susceptibility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Individuals with high risk for Alzheimer's disease
  Interventions: Procedure: BOLD and Perfusion brain MRI
- 2: Individuals with low risk for Alzheimer's disease
  Interventions: Procedure: BOLD and Perfusion brain MRI

INTERVENTIONS:
Procedure: BOLD and Perfusion brain MRI — Blood oxygenation and perfusion functional MRI performed twice, two weeks apart; each scan lasts 1 hour

SUMMARY:
The purpose of this study is to develop imaging techniques that can distinguish functional brain changes in people at high risk for dementia years prior to onset of clinical memory problems from those with normal changes of aging.

DETAILED DESCRIPTION:
The overall goals of this project are to identify consistent patterns of variance in brain function in patients at risk for Alzheimer's Disease by using APOE ε4 as a marker for disease risk. The activation Blood Oxygen Level Dependency (BOLD) signal will be compared to both resting and activation perfusion signals to assess the variability of cerebral blood flow as it relates to the BOLD signal. Each participant will be imaged on a 3T MRI scanner while performing an associate episodic memory task.

A total of 90 individuals will be recruited for this study. Participants will be non-demented, right handed, adults with or without at least one APOE ε4 allele. Groups will be split as follows: A) ages 25-39: non-ε4 (n=15); B) ages 25-39: +ε4 (n=15); C) ages 40-49: non-ε4 (n=15); D) ages 40-49: +ε4 (n=15);.E) ages 50-65: non-ε4: F) ages 50-65: +ε4 (n=15). These groups will be matched for mean age, mean years of education, gender distribution, as well as the presence or absence of a family history of AD in a first degree relative.

There will be 2 scanning sessions for each participant. Scan session #1 and Scan session #2 will be acquired within 2 weeks of each other and will take approximately one hour each.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed

Exclusion Criteria:

* Major medical illnesses
* History of significant head trauma with residual cognitive deficits
* Other neurological or major psychiatric disorders such as schizophrenia, bipolar disorder, developmental learning disorder, and alcohol or substance abuse
* MRI contra-indications

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy adults from the community
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2005-08; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
identification of consistent patterns of variance in brain function in subjects at risk for Alzheimer's Disease by using APOE ε4 as a marker for disease risk | single time point

CONTACTS AND LOCATIONS:
Overall Officials: Adam Fleisher, MD, Principal Investigator — University of California, San Diego
Locations (1):
- Shiley-Marcos Alzheimer's Disease Research Center, University of California, San Diego, La Jolla, California, United States

REFERENCES:
- [Background] Bookheimer SY, Strojwas MH, Cohen MS, Saunders AM, Pericak-Vance MA, Mazziotta JC, Small GW. Patterns of brain activation in people at risk for Alzheimer's disease. N Engl J Med. 2000 Aug 17;343(7):450-6. doi: 10.1056/NEJM200008173430701. PMID 10944562
- [Background] Mayeux R, Ottman R, Tang MX, Noboa-Bauza L, Marder K, Gurland B, Stern Y. Genetic susceptibility and head injury as risk factors for Alzheimer's disease among community-dwelling elderly persons and their first-degree relatives. Ann Neurol. 1993 May;33(5):494-501. doi: 10.1002/ana.410330513. PMID 8498827
- [Background] Fleisher AS, Houston WS, Eyler LT, Frye S, Jenkins C, Thal LJ, Bondi MW. Identification of Alzheimer disease risk by functional magnetic resonance imaging. Arch Neurol. 2005 Dec;62(12):1881-8. doi: 10.1001/archneur.62.12.1881. PMID 16344346
- [Background] Fleisher A, Grundman M, Jack CR Jr, Petersen RC, Taylor C, Kim HT, Schiller DH, Bagwell V, Sencakova D, Weiner MF, DeCarli C, DeKosky ST, van Dyck CH, Thal LJ; Alzheimer's Disease Cooperative Study. Sex, apolipoprotein E epsilon 4 status, and hippocampal volume in mild cognitive impairment. Arch Neurol. 2005 Jun;62(6):953-7. doi: 10.1001/archneur.62.6.953. PMID 15956166